CLINICAL TRIAL: NCT00154791
Title: Phase I/II Trial of Biweekly Gemcitabine, Oxaliplatin, and 48-Hour Infusion of High-Dose 5-FU/Leucovorin (GOFL) in Advanced Pancreatic Adenocarcinoma
Brief Title: Phase I/II Trial GOFL in Advanced Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 900905
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-08

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; Oxaliplatin; Gemcitabine; 5-FU
MeSH Terms: interventions — Oxaliplatin; Gemcitabine

INTERVENTIONS:
Drug: oxaliplatin
Drug: gemcitabine
Drug: 5-FU/LV

SUMMARY:
We plan to conduct a phase I/II clinical trial using biweekly gemcitabine, oxaliplatin, and 48-hour infusion of high dose 5-FU/leucovorin to treat patients with advanced pancreatic adenocarcinoma. In the phase I part, the maximum tolerable dose of oxaliplatin in combination with biweekly gemcitabine 800 mg/m2 and 48-hour infusion of 5-FU 3000 mg/m2 and leucovorin 300 mg/m2 will be determined. In the phase II part, the efficacy and safety of the biweekly chemotherapy with GOFL will be evaluated.

DETAILED DESCRIPTION:
For each dose of GOFL chemotherapy, intravenous infusion of gemcitabine at a fixed rate of 10 mg/m2/min will be immediately followed by a 2-hour intravenous infusion of oxaliplatin and then a 48-hour intravenous infusion of 5-FU and leucovorin.The starting dose of oxaliplatin in the phase I part is 65 mg/m2, with dose increment of 10 mg/m2. Since the recommended dose for biweekly single dose oxaliplatin is 85 mg/m2, there will be no further dose escalation of oxaliplatin beyond 85 mg/m2.Patients will be entered in cohorts of three.If one out of three patients develops DLT, three additional patients will be accrued to the same dose level.9.1.3 The six patients treated at the MTD dose level will be included in the phase II part of this study if only they have measurable lesion(s) prior to chemotherapy.For the phase II part, If three or more responders are observed in the initial 21 evaluable patients, the trial will proceed to the second stage. Additional 24 patients will be accrued in the second stage of the phase II part.

ELIGIBILITY:
Inclusion Criteria:

* 5.1.1 Patients must have metastatic or unresectable adenocarcinoma of the pancreas. The diagnosis of pancreatic adenocarcinoma must be confirmed by histopathology or cytology.

5.1.2 For the phase I part of this trial, patients who have disease measurable or evaluable on x-ray, CAT scan, or physical examination are eligible. For the phase II part of this trial, only patients who have disease measurable on x-ray, CAT scan, or physical examination are eligible.

5.1.3 Patients must have no history of prior chemotherapy. 5.1.4 Patients with prior radiotherapy are eligible if the irradiated area is not the only source of measurable or evaluable disease.

5.1.5 Patients' baseline ECOG performance status must be £ 2. 5.1.6 Patients' life expectancy must be 12 weeks or greater. 5.1.7 Patients' age must be ³ 20 and £ 75. 5.1.8 Patients must have adequate bone marrow function, defined as WBC count ³ 3,500/ul, neutrophil count ³ 1,500/ul, and platelet count ³ 100,000/ul.

5.1.9 Patients must have adequate liver function and adequate renal function, defined as the following: serum alanine (ALT) £ 5 times upper normal limit, serum total bilirubin level £ 2.0 mg/dL, and serum creatinine £ 1.5 mg/dL.

5.1.10 Patients who have biliary obstruction and have undergone adequate drainage procedures before enrollment are eligible.

5.1.11 Patients must agree to have indwelling venous catheter implanted. 5.1.12 Women or men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

5.1.13 All patients must be informed of the investigational nature of this study and must sign and give written informed consent.

Exclusion Criteria:5.2.1 Patients who have central nervous system metastasis 5.2.2 Patients who have active infection 5.2.3 Pregnant or breast-nursing women 5.2.4 Patients who have active cardiac disease or history of ischemic heart disease 5.2.5 Patients who have peripheral neuropathy > Grade I of any etiology 5.2.6 Patients who have serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator) 5.2.7 Patients who have other prior or concurrent malignancy except for adequately treated in situ carcinoma of cervix or adequately treated basal cell carcinoma of skin 5.2.8 Patients who are under biologic treatment for their malignancy

-

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2003-03; Study Completion 2005-08

PRIMARY OUTCOMES:
Primary objective: to evaluate the maximum tolerated dose of oxaliplatin in phase I part and to evaluate the objective tumor response rate of GOFL in phase II part

SECONDARY OUTCOMES:
To evaluate clinical benefit response, overall survival of GOFL

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D.Ph.D, Study Chair — National Health Research Institutes, Division of Cancer Research; Hui-Ju Ch'ang, M.D., Principal Investigator — National Taiwan University Hospital; Chih-Hung, Hsu, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan